CLINICAL TRIAL: NCT06326450
Title: Remote Augmented Reality Versus Traditional In-person Resuscitation Assessment: an International Noninferiority Randomized Controlled Trial
Brief Title: Traditional In-Person Vs. Remote AR Clinical Simulation
Acronym: AR Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 74626
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Educational Problems
Keywords: Augmented Reality; Advanced Cardiac Life Support; Clinical Simulation; Medical Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Augmented Reality Enhanced Simulation (Treatment group) (Experimental): Participants will experience augmented simulations with a holographic mixed-reality setting based on different workplace scenarios such as medical crisis via Augmented Reality (AR) headset.
  Interventions: Behavioral: Augmented Reality simulation
- Traditional In Situ Simulation (Control group) (Active Comparator): Participants will experience in-person simulations of different workplace scenarios such as medical error and workplace harassment
  Interventions: Behavioral: In Person simulation

INTERVENTIONS:
Behavioral: Augmented Reality simulation — Augmented simulation of medical crisis scenarios
  Arms: Experimental: Augmented Reality Enhanced Simulation (Treatment group)
Behavioral: In Person simulation — In Person simulation of medical crisis scenarios
  Arms: Traditional In Situ Simulation (Control group)

SUMMARY:
This is a non-inferiority, international, controlled trial that aims to evaluate the progression of physicians and residents through an Advanced Cardiac Life Support (ACLS) clinical simulated scenario. The study's primary objective is to compare the performance outcomes between two groups: participants in the traditional in-person simulation and those immersed in the Augmented Reality (AR) scenario

ELIGIBILITY:
Inclusion Criteria:

* Brazilian resident

Exclusion Criteria:

* a history of severe motion sickness
* currently have nausea
* a history of seizures
* wear corrective glasses.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-06-22 (Actual); Primary Completion 2024-08-03 (Actual); Study Completion 2024-08-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of Technical Skill (TS) and Non Technical Skill (NTS) Performance | immediately after simulation
  Measured with Instrument for the evaluation of advanced life support performance. The instrument consists of 26 items, which are rated on a scale from +2 to -2. A total assessment score of performance is given based on a scale from 0 to 10 (0=poor, 10=excellent) at the end of the instrument.

SECONDARY OUTCOMES:
Reassessment of Non Technical Skill (NTS) with Behaviorally Anchored Rating Scale (BARS) | immediately after simulation
  Measured with individual Behaviorally Anchored Rating Scale (BARS). The BARS scoring system uses four categories assessing situation awareness, decision-making, communication and teamwork. The score ranges from 1 and 9 (1 = poor and 9 = excellent)
Evaluation of the AR system's usability | immediately after simulation
  Measured with the System Usability Scale (SUS). The scale has 10 items. Scores ranges from 1-5 (1 = strongly disagree and 5 = strongly agree)
Evaluation of the AR system's ergonomics | immediately after simulation
  Measured with the ISO 9241-400 Assessment of human-ergonomic factors. The scale has 6 items. Scores ranges from 1-5 (1 = strongly disagree and 5 = strongly agree)

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Parkard Children's Hospital, Stanford, California, United States